CLINICAL TRIAL: NCT02490592
Title: Comparison of the Effect of Fluoride Remineralizer Gel and Foam: a Randomized Clinical Trial
Brief Title: Comparison of the Effect of Fluoride Remineralizer Gel and Foam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Center of João Pessoa (Other)
Collaborators: Universidade Cruzeiro do Sul (Other)
Responsible Party: Principal Investigator, JAINARA MARIA SOARES FERREIRA, JAINARA MARIA SOARES FERREIRA, University Center of João Pessoa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAAE: 25687413.8.000.5176
Record Dates: First submitted 2014-10-28; First posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G1 (Experimental): Thirty children aged seven to twelve years who had seventy one active white spots lesions in permanent anterior teeth randomly assigned to four or eight weekly intervals applications of fluoride foam, Flúor Care (NaF 1.23%), to verified the activity (visual scores) and the dimensional changes of whit spot lesions (with WHO probe and millimeter ruler), caries Management by Risk Assessment (CAMBRA) and OHI-S (Simplified Oral Hygiene Index) of children.
  Interventions: Other: Fluoride Foam
- G2 (Experimental): Twenty-eight children aged seven to twelve years who had seventy five active white spots lesions in permanent anterior teeth randomly assigned to four or eight weekly intervals applications of fluoride gel, Flugel FFA (NaF 1.23%), to verified the activity (visual scores) and the dimensional changes of whit spot lesions (with WHO probe and millimeter ruler), caries Management by Risk Assessment (CAMBRA) and OHI-S (Simplified Oral Hygiene Index) of children.
  Interventions: Other: Fluoride gel

INTERVENTIONS:
Other: Fluoride Foam — Fluoride foam - Flúor Care (NaF 1.23%) (G1)
  Arms: G1
Other: Fluoride gel — Fluoride gel - Flugel FFA (NaF 1.23%) (G2)
  Arms: G2

SUMMARY:
Compare the remineralizing effect of acidulated fluoride gel Flugel (1.23% FFA, DFL) and acidulated Fluoride Foam Flúor Care (1.23% FFA, FGM) in maxillary anterior permanent teeth of 58 children aged 7 to 12 years of age.

to verified the activity (visual scores) and the dimensional changes of whit spot lesions (with WHO probe and millimeter ruler), risk for caries (CAMBRA) and OHI-S (Simplified Oral Hygiene Index) of children.

DETAILED DESCRIPTION:
This randomized clinical trial was composed permantentes previous teeth with white spot esolares belonging to the age group 7-12 years of the interior of Paraíba (Brazil). To calculate the sample considered the study of Soares and Valencia (2003) who obtained success rate of inactivity for white patches of fluoride gel (41%) compared with fluoride varnish (33%). By means of the Epi Info program™ 6 was used maximum acceptable error α and β of 5% to 20% ratio equal to 1.0 between the two products, resulting in a representative sample of 47 cases for each group for a total 94 white spots. To account for any loss sample, the sample was extended to 146 white spots being the case 71 formed by G1 and G2 for 75 cases. Prior to implementation of the proposed study called a calibration INLUX through 46 images of white spots followed by the investigation of the reproducibility of tests using Kappa coefficient intra and inter examiner with 10% of the sample (n = 14) was performed. The interpretation of these statistical testing was performed according to scale Bulman and Osborn (1989). There was a correlation of intra k = 1.00 (good) activity for k = 1.00 (good) scale for all considered good. Already on inter-examiner agreement, the investigators observed values of k = 1.00 (good) for activity k = 0.65 (substantial) for dimension being considered, good and substantial, respectively. For this study the investigators followed the following protocol: the IHO S-Record (Simplified Oral Hygiene Index); Supervised brushing; Professional prophylaxis; drying; Evaluation of white spot (the enamel was visually assessed at the initial examination (S1), after the 4th (S5) and 8th (S9) weeks of fluoride products only stains that were not remineralized to S5, the activity (visual scores by Nyvad et al (1999)) and the dimensional changes (with WHO probe and millimeter ruler); Caries Management by Risk Assessment (CAMBRA); Application of fluoride products: group 1 (G1) where children received weekly therapeutic applications of fluoridated foam FFA, Flúor Care (NaF 1.23%) or group 2 (G2) where children received applications weekly therapeutic fluoride gel Flugel FFA (1.23% NaF) the management of this study was performed according to the CONSORT (Consolidated Standards of ReportingTrials) your flowchart comprises four stages of a controlled clinical trial:. recruitment, allocation, follow-up . analysis and the project was approved by the ethics committee in Brazil on February 27, 2014 (CAAE: 25687413.8.000.5176).

ELIGIBILITY:
Inclusion Criteria:

* Child with active incipient caries lesions (white spots) on upper anterior permanent teeth; permission from parents / guardians through the consent form, authorization of the minor through the term of assent, children at high risk for dental caries.

Exclusion Criteria:

* Children who used braces, medications that alter the flow / salivary composition or antibiotics in the month before the exam. Not patients with syndromes or changes in tooth development, patients with cognitive and motor disorders were included.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
visual scores | within the first 60 days
  activity changes of whit spot lesions
millimeters (with WHO probe and millimeter ruler) | within the first 60 days
  dimensional changes of whit spot lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jainara Ferreira, Phd, Principal Investigator — UNIPÊ